CLINICAL TRIAL: NCT06838533
Title: Patient Specific Polyetheretherketone (PEEK) Miniplates Versus Titanium Genioplasty Plates in The Fixation of Computer-Guided Advancement Genioplasty
Brief Title: Patient Specific PEEK Versus Titanium Patient Specific Plates in The Fixation of Computer-Guided Advancement Genioplasty
Acronym: PEEK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Principal Investigator, Dina Mohamed Mohamed Abdelwahab, Principal Investigator, Faculty of Dental Medicine for Girls
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORSUR-108-2-L
Record Dates: First submitted 2025-02-12; First posted 2025-02-20 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Mandible; Deformity
Keywords: Genioplasty; PEEK; Mandible deformity
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEEK plates in Computer guided advancement genioplasty (Experimental): Study group
  Interventions: Procedure: computer guided advancement genioplasty
- Titanium plates in Computer guided advancement genioplasty (Experimental): Control group
  Interventions: Procedure: computer guided advancement genioplasty

INTERVENTIONS:
Procedure: computer guided advancement genioplasty — PEEK vs Titanium patient specific plates

SUMMARY:
Evaluation of polyetheretherketone (PEEK) versus titanium patient specific plates in the fixation of computer-guided advancement genioplasty.

DETAILED DESCRIPTION:
Aim: Comparison between polyetheretherketone (PEEK) and titanium patient specific plates in the fixation of computer-guided advancement genioplasty.

Patients and Methods: This study included fourteen patients indicated for advancement genioplasty. Patients were assigned randomly into one of two equal groups. Group A (Control group) included seven patients who were treated by computer guided advancement genioplasty using patient specific titanium plates and Group B(Study group) involved seven patients who were treated by computer guided advancement genioplasty using patient specific PEEK plates.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are indicated to advancement genioplasty.
* Patients with completed growth.
* Physically and psychologically able to tolerate surgical procedures.

Exclusion Criteria:

* Presence of any medical conditions that contraindicate the surgical procedure.
* Any medical condition that compromises the healing and surgical outcome.

Ages: 17 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2018-03-03 (Actual); Primary Completion 2024-03-02 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Stability of PEEK vs Titanium plates | 6 months follow up
  Radiographic linear discrepancy in mm (Horizontal and vertical) between Pogonion and Menton position in immediate and 6 months postoperative

SECONDARY OUTCOMES:
Patient satisfaction | 6 months
  Number from 1 to 5 of a 5-point Likert scale (1 very dissatisfied is minimal to 5 very satisfied is maximum)
Cost of patient specific plated (PEEK and titanium) | 6 months
  Number in Egyptian pound
Soft tissue healing | 6 months
  Binary answer (yes if happened or no if not happened) of clinical examination (Infection, soft tissue dehiscence and plate exposure)

CONTACTS AND LOCATIONS:
Overall Officials: Nahed Adly, consultant, Study Director — Assistant professor at faaculty of dentistry AlAzhar university
Locations (1):
- Dina mohamed abdelwahab, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/33/NCT06838533/Prot_SAP_ICF_000.pdf